CLINICAL TRIAL: NCT06137027
Title: Sublingual Cannabidiol Oil Extract for Prevention of Postoperative Nausea and Vomiting in Elective Gynaecological Patients at the University Hospital of the West Indies (UHWI)
Brief Title: Cannabidiol Oil Extract for Prevention of Postoperative Nausea and Vomiting
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CREC-MN.0722/2022/2023
Record Dates: First submitted 2023-05-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Cannabidiol oil; Postoperative nausea and vomiting; Patient satisfaction
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Patient Satisfaction | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: The intervention group will receive Cannabidiol oil 5.5mg sublingually (10 drops). The control group will receive a peppermint based oil sublingually (10 drops).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, researcher administering the agent and the attending anaesthetist will all be blinded to the agent administered. Only the pharmacist preparing the oil will know what it contains.
  Patients will be allocated into one of two groups:
  Group 1 - Intervention group Group 2 - Placebo group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol Oil (Active Comparator): Cannabidiol oil 5.5mg, equivalent to 10 drops
  Interventions: Drug: Cannabidiol Oil
- Placebo (Placebo Comparator): Peppermint oil, 10 drops
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol Oil — Cannabidiol oil will be administered sublingually 2-3 hours preoperatively
  Other Names: CBD
  Arms: Cannabidiol Oil
Drug: Placebo — Placebo will be administered sublingually 2-3 hours preoperatively
  Other Names: PLA
  Arms: Placebo

SUMMARY:
Cannabidiol oil has been shown to be effective in treating chemotherapy induced nausea and vomiting, but there is limited information on its usefulness in nausea and vomiting that can occur after surgery. The goal of this study is to determine the effect of Cannabidiol oil on the frequency of nausea and vomiting in the first 24 hours after a gynaecological procedure. Other effects that will be assessed will include:

1. The effect of Cannabidiol oil on the level of pain and amount of pain medications needed in the first 24 hours after a gynaecological operation.
2. The effect of Cannabidiol oil on patients' overall satisfaction with the anaesthetic experience.

Some participants will be administered Cannabidiol oil under the tongue two to three hours before their procedure and an equal number will receive a placebo oil, similar in taste. This will be done randomly to minimise introducing bias. We will then compare both groups in the postoperative period to see if the Cannabidiol oil made any difference.

DETAILED DESCRIPTION:
The overall aim of this study is to evaluate the effect of Cannabidiol oil on postoperative nausea and vomiting in elective gynaecological surgical patients undergoing general anaesthesia at the University Hospital of the West Indies, Jamaica and to determine if total analgesic requirements are reduced in the intervention group in the first 24 hours.

Primary Objective:

To compare the incidence of postoperative nausea and vomiting in gynaecological patients who receive 5.5mg of Cannabidiol oil sublingually two to three hours preoperatively to those receiving a placebo in adult elective gynaecological surgical patients.

Secondary Objectives:

* To compare the total amount of rescue anti-emetic medications administered in the first 24 hours postoperatively between the group receiving Cannabidiol oil and the placebo group.
* To compare total analgesic requirements in the first 24 hours postoperatively between those receiving Cannabidiol oil and the placebo group.
* To compare the level of patient satisfaction with the overall anaesthetic experience between the intervention group and the placebo group.

We propose to use a dose of 5.5mg sublingually based on studies which have demonstrated the effectiveness of these for chemotherapy induced vomiting. As there are numerous factors which may affect postoperative nausea and vomiting, including sex, type of surgery and degree of postoperative pain, we will include only female patients undergoing gynaecological surgery to minimise these confounding factors. Of note, this patient group is one of the high-risk groups for postoperative nausea and vomiting, with an incidence in obstetrics and gynaecology of 40-80%. Cannabidiol oil is typically well tolerated with a favourable side effect profile as it non psychoactive. Previous studies have documented that the most common side effects observed were somnolence, sedation and altered mood.

Recruitment of patients will be done on the ward on the day prior to surgery. Time will be allowed for questioning and gathering of information and all risks will be explained. Written consent will be obtained by the researcher, or the research assistant, who will not be involved in the intra-operative management of the patient. The preoperative assessment will be conducted by the anaesthetist as per usual.

The study will be a single centre, double-blinded (patient and attending Anaesthetist) randomised controlled trial. Patients will be randomly allocated into one of two groups:

* Group 1 - Intervention group
* Group 2 - Placebo group

A sample size of 120 patients was calculated, 60 per group, based on an alpha value of 0.05, beta value of 0.2 and an expected proportion of 50%. An increase by 10% was done to address anticipated drop outs. The Intervention group will receive 5.5mg (10 drops) of Cannabidiol oil (infused peppermint oil) sublingually. The placebo group will receive 10 drops of peppermint oil or similar taste.

The intervention (Cannabidiol oil) and placebo will be placed in identical amber, 2ml glass bottles, each having a different assigned number-letter code. The assigned codes will be computer generated and the bottles will be labelled by the pharmacist. The participants will be randomised using an online randomiser programme (www.randomization.com). The pharmacist will assign an appropriate code to the patient/s based on the randomisation table on the day prior to surgery, which will be given to the researcher.

Two to three hours prior to surgery, the assigned agent will be administered by the researcher or assistant. The person administering the intervention will not participate in the conduct of anaesthesia or the collection of data. A protocol is in place to monitor and manage any untoward adverse drug reactions, including anaphylaxis. A standardized technique of General Anaesthesia will be implemented:

* Induction with propofol at 2mg/kg
* Muscle relaxation with Cisatracurium 0.1mg/kg
* Morphine 0.1mg/kg
* Panadol 1g

Data will be collected on medications administered, length of anaesthesia and estimated blood loss. For antiemetic prophylaxis, a standardised protocol of dexamethasone 8mg and dimenhydrinate 0.5mg/kg (~50mg) will be given. In the postoperative period, the rescue protocol in the event of an episode of vomiting or severe nausea is as follows:

1. Step 1: Repeat dose of dexamethasone 4mg
2. Step 2 if no resolution: Kytril 1mg

The proposed study will also include an assessment of the risk of post operative nausea and vomiting, assessment of the presence and severity of any nausea and vomiting and an assessment of patient satisfaction with their overall anaesthesia experience. The Apfel score will be used to assess the risk of postoperative nausea and vomiting, and includes four factors: sex, smoking history, previous history of nausea and vomiting or motion sickness and any plan to use postoperative opioids by the medical team. This produces a score between I and IV and the risk of postoperative nausea and vomiting increases with an increasing score. An Apfel score of I usually carries a 20% risk of postoperative nausea and vomiting and this increases to 80% with a score of IV. The purpose of determining the Apfel score at the time of written consent is to evaluate the effect of the Cannabidiol intervention on not only the overall incidence of postoperative nausea and vomiting, but also to be able to determine how it affects different risk groups. The BARF scale will be used to assess the presence of nausea, which is a subjective sensation and challenging to capture.It consists of six faces, with a scale from 0 to 10. The BARF scale will be checked on arrival to and on discharge from the Post Anaesthetic Care Unit. The Leiden Peri-operative care Patient Satisfaction questionnaire (LPPSq) will be used to assess patient satisfaction and will be conducted 24 to 48 hours postoperatively. It assesses satisfaction with respect to information received, any fears and concerns, professional competence, service and staff-patient relationships.

The data will be collected by the anaesthesia and recovery room nursing staff from the intra-operative anaesthetic and recovery room records. The researcher will then collect all sheets and conduct the patient satisfaction questionnaire between 24 and 48 hours postoperatively. The Apfel score will be assessed by the anaesthetist in charge of the patient at the preoperative visit. The BARF scale will be done by the recovery room and ward nursing staff.

Data will be entered into and analysed using SPSS v. 26.

ELIGIBILITY:
Inclusion Criteria:

All patients for elective gynaecological surgical procedures under general anaesthesia at the Main operating theatre, UHWI between the ages of 18-65 years.

Exclusion Criteria:

* Reported allergy to cannabis/CBD by products, coconut oil, peppermint oil
* Patients < 18 years
* Patients experiencing disease related nausea and vomiting
* Patients with psychological/psychiatric illnesses which prevent communication or impairs their ability to give informed consent
* Patients undergoing regional anaesthesia
* Contraindication to medicinal cannabis such as unstable cardiovascular disease, substance use disorder, or significant mental health disorder
* Cannabis use within 30 days of surgery
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Post Operative Vomiting | 24 hours post surgery
  All episodes of vomiting will be recorded by the nursing staff in the Post anaesthesia care unit and after discharge, by the ward nurses for the first 24 hours after surgery.
Postoperative Nausea | 24 hours post surgery
  The BARF score will be administered by the nursing staff in the Post anaesthesia care unit to assess nausea on admission and on discharge from the unit. It will also be assessed by the ward nurses at 4 hour intervals during vital checks for the first 24 hours after surgery.

SECONDARY OUTCOMES:
Total analgesic requirements | 24 hours post surgery
  All analgesics administered in the Post Anaesthesia Care unit and on the ward up to 24 hours post procedure will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Tennant, DM, PhD, Principal Investigator — University Hospital of the West Indies
Locations (1):
- University Hospital of the West Indies, Kingston, Jamaica

REFERENCES:
- [Background] Becker DE. Nausea, vomiting, and hiccups: a review of mechanisms and treatment. Anesth Prog. 2010 Winter;57(4):150-6; quiz 157. doi: 10.2344/0003-3006-57.4.150. PMID 21174569
- [Background] Bashashati M, McCallum RW. Neurochemical mechanisms and pharmacologic strategies in managing nausea and vomiting related to cyclic vomiting syndrome and other gastrointestinal disorders. Eur J Pharmacol. 2014 Jan 5;722:79-94. doi: 10.1016/j.ejphar.2013.09.075. Epub 2013 Oct 22. PMID 24161560
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Kakodkar PS. Routine use of dexamethasone for postoperative nausea and vomiting: the case for. Anaesthesia. 2013 Sep;68(9):889-91. doi: 10.1111/anae.12308. Epub 2013 Jul 15. No abstract available. PMID 23848292
- [Background] Tien M, Gan TJ, Dhakal I, White WD, Olufolabi AJ, Fink R, Mishriky BM, Lacassie HJ, Habib AS. The effect of anti-emetic doses of dexamethasone on postoperative blood glucose levels in non-diabetic and diabetic patients: a prospective randomised controlled study. Anaesthesia. 2016 Sep;71(9):1037-43. doi: 10.1111/anae.13544. PMID 27523051
- [Background] Roden DM. Drug-induced prolongation of the QT interval. N Engl J Med. 2004 Mar 4;350(10):1013-22. doi: 10.1056/NEJMra032426. No abstract available. PMID 14999113
- [Background] Kothari SN, Boyd WC, Bottcher ML, Lambert PJ. Antiemetic efficacy of prophylactic dimenhydrinate (Dramamine) vs ondansetron (Zofran): a randomized, prospective trial inpatients undergoing laparoscopic cholecystectomy. Surg Endosc. 2000 Oct;14(10):926-9. doi: 10.1007/s004640080055. PMID 11080405
- [Background] Cabral GA, Raborn ES, Griffin L, Dennis J, Marciano-Cabral F. CB2 receptors in the brain: role in central immune function. Br J Pharmacol. 2008 Jan;153(2):240-51. doi: 10.1038/sj.bjp.0707584. Epub 2007 Nov 26. PMID 18037916
- [Background] D'Souza DC, Perry E, MacDougall L, Ammerman Y, Cooper T, Wu YT, Braley G, Gueorguieva R, Krystal JH. The psychotomimetic effects of intravenous delta-9-tetrahydrocannabinol in healthy individuals: implications for psychosis. Neuropsychopharmacology. 2004 Aug;29(8):1558-72. doi: 10.1038/sj.npp.1300496. PMID 15173844
- [Background] Parker LA, Rock EM, Limebeer CL. Regulation of nausea and vomiting by cannabinoids. Br J Pharmacol. 2011 Aug;163(7):1411-22. doi: 10.1111/j.1476-5381.2010.01176.x. PMID 21175589
- [Background] Legare CA, Raup-Konsavage WM, Vrana KE. Therapeutic Potential of Cannabis, Cannabidiol, and Cannabinoid-Based Pharmaceuticals. Pharmacology. 2022;107(3-4):131-149. doi: 10.1159/000521683. Epub 2022 Jan 28. PMID 35093949
- [Background] Izzo AA, Borrelli F, Capasso R, Di Marzo V, Mechoulam R. Non-psychotropic plant cannabinoids: new therapeutic opportunities from an ancient herb. Trends Pharmacol Sci. 2009 Oct;30(10):515-27. doi: 10.1016/j.tips.2009.07.006. Epub 2009 Sep 2. PMID 19729208
- [Background] Grimison P, Mersiades A, Kirby A, Lintzeris N, Morton R, Haber P, Olver I, Walsh A, McGregor I, Cheung Y, Tognela A, Hahn C, Briscoe K, Aghmesheh M, Fox P, Abdi E, Clarke S, Della-Fiorentina S, Shannon J, Gedye C, Begbie S, Simes J, Stockler M. Oral THC:CBD cannabis extract for refractory chemotherapy-induced nausea and vomiting: a randomised, placebo-controlled, phase II crossover trial. Ann Oncol. 2020 Nov;31(11):1553-1560. doi: 10.1016/j.annonc.2020.07.020. Epub 2020 Aug 13. PMID 32801017
- [Background] Hosseini A, McLachlan AJ, Lickliter JD. A phase I trial of the safety, tolerability and pharmacokinetics of cannabidiol administered as single-dose oil solution and single and multiple doses of a sublingual wafer in healthy volunteers. Br J Clin Pharmacol. 2021 Apr;87(4):2070-2077. doi: 10.1111/bcp.14617. Epub 2020 Nov 18. PMID 33075170
- [Background] Nitecka-Buchta A, Nowak-Wachol A, Wachol K, Walczynska-Dragon K, Olczyk P, Batoryna O, Kempa W, Baron S. Myorelaxant Effect of Transdermal Cannabidiol Application in Patients with TMD: A Randomized, Double-Blind Trial. J Clin Med. 2019 Nov 6;8(11):1886. doi: 10.3390/jcm8111886. PMID 31698733
- [Background] Alaia MJ, Hurley ET, Vasavada K, Markus DH, Britton B, Gonzalez-Lomas G, Rokito AS, Jazrawi LM, Kaplan K. Buccally Absorbed Cannabidiol Shows Significantly Superior Pain Control and Improved Satisfaction Immediately After Arthroscopic Rotator Cuff Repair: A Placebo-Controlled, Double-Blinded, Randomized Trial. Am J Sports Med. 2022 Sep;50(11):3056-3063. doi: 10.1177/03635465221109573. Epub 2022 Jul 29. PMID 35905305
- [Background] Echeverria-Villalobos M, Fiorda-Diaz J, Uribe A, Bergese SD. Postoperative Nausea and Vomiting in Female Patients Undergoing Breast and Gynecological Surgery: A Narrative Review of Risk Factors and Prophylaxis. Front Med (Lausanne). 2022 Jul 1;9:909982. doi: 10.3389/fmed.2022.909982. eCollection 2022. PMID 35847822
- [Background] Mahmood L, Hegde R, Mariswami M, Ollapally A. Validation of the Apfel scoring system for identification of High-risk patients for PONV. Karnataka Anaesthesia Journal. 2015;1:115.
- [Background] White P, Shafer A, editors. Nausea and vomiting: causes and prophylaxis. Seminars in anesthesia; 1987
- [Background] Baxter AL, Watcha MF, Baxter WV, Leong T, Wyatt MM. Development and validation of a pictorial nausea rating scale for children. Pediatrics. 2011 Jun;127(6):e1542-9. doi: 10.1542/peds.2010-1410. Epub 2011 May 29. PMID 21624874
- [Background] Şişman H, Aslan F, Özgen R, Alptekin D, Akil Y. Validity and Reliability Study of the Baxter Animated Retching Faces Nausea Scale. Journal of Pediatric Surgical Nursing. 2016;5:98-106.
- [Background] Caljouw MA, van Beuzekom M, Boer F. Patient's satisfaction with perioperative care: development, validation, and application of a questionnaire. Br J Anaesth. 2008 May;100(5):637-44. doi: 10.1093/bja/aen034. Epub 2008 Mar 12. PMID 18337271
- [Background] Jlala HA, Caljouw MA, Bedforth NM, Hardman JG. Patient satisfaction with perioperative care among patients having orthopedic surgery in a university hospital. Local Reg Anesth. 2010;3:49-55. doi: 10.2147/lra.s11381. Epub 2010 Jul 28. PMID 22915869